CLINICAL TRIAL: NCT00911560
Title: Phase I/II Trial of a Bivalent Vaccine With Escalating Doses of the Immunological Adjuvant OPT-821, in Combination With Oral β-glucan for High-Risk Neuroblastoma
Brief Title: Bivalent Vaccine With Escalating Doses of the Immunological Adjuvant OPT-821, in Combination With Oral β-glucan for High-Risk Neuroblastoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 05-075
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Neuroblastoma
Keywords: BETA-D-GLUCAN; OPT-821; GD2-KLH; GD3-KLH; QS 21; Vaccine; 05-075
MeSH Terms: conditions — Neuroblastoma

ARMS (3):
- vaccine group one (Experimental): Patients will receive a total of 7 subcutaneous injections, at weeks 1, 2, 3, 8 , 20 , 32 , and 52. Minor schedule adjus tment s are permitted , as needed Vaccines must occur a inimum of 6 days apart. The last three vaccine s can be administered up to one week earlier or later than indicated without representing a protocol violation.Patients assigned to in Group 1 will receive o ral β glucan (40 mg/kg/day) starting at week 6 or 7 and continue with approximately 2 weeks on, 2 weeks off, up to 1 cycle after the last vaccination .
  Interventions: Biological: adjuvant OPT-821 in a vaccine containing two antigens (GD2L and GD3L) covalently linked to KLH; Biological: oral β-glucan
- vaccine group two (Experimental): Patients will receive a total of 7 subcutaneous injections, at weeks 1, 2, 3, 8 , 20 , 32 , and 52. Minor schedule adjus tment s are permitted , as needed Vaccines must occur a minimum of 6 days apart. The last three vaccine s can be administered up to one week earlier or later than indicated without representing a protocol violation.Patients assigned to Group 2 will receive oral β glucan (40 mg/kg/day) starting week 1 and continue with approximately 2 weeks on, 2 weeks off, up to 1 cycle after the last vaccination .
  Interventions: Biological: adjuvant OPT-821 in a vaccine containing two antigens (GD2L and GD3L) covalently linked to KLH; Biological: oral β-glucan
- vaccine group three (Experimental): Patients will receive a total of 7 subcutaneous injections, at weeks 1, 2, 3, 8 , 20 , 32 , and 52. Minor schedule adjus tment s are permitted , as needed Vaccines must occur a minimum of 6 days apart. The last three vaccine s can be administered up to one week earlier or later than indicated without representing a protocol violation.Group 3 will include patients who have previously received vaccine and oral β glucanglucan. Patients in this group will not be randomized using the MSK CRDB system. They will be treated as patients in Group 1 and receive o ral β glucan (40 mg/kg/day) starting at week 6 or 7 and continue with approximately 2 weeks on, 2 weeks off, up to 1 cycle after the last vaccination . They will not be eligible for primary endpoint.
  Interventions: Biological: adjuvant OPT-821 in a vaccine containing two antigens (GD2L and GD3L) covalently linked to KLH; Biological: oral β-glucan

INTERVENTIONS:
Biological: adjuvant OPT-821 in a vaccine containing two antigens (GD2L and GD3L) covalently linked to KLH — Pts receive a total of 7 subcutaneous injections, at weeks 1, 2, 3, 8, 20, 32, & 52. Minor schedule adjustments are permitted, as needed. Vaccines must occur a minimum of 6 days apart. Induction of antibody response against the target antigens will be assessed. A fixed dose of oral β-glucan (40 mg/kg/day) is started at week 6 or 7(to allow time for generation of antibodies), & continued as approximately 2 weeks on, 2 weeks off, up to 1 cycle after the last vaccination. Neutrophils will be tested for glucan effects on cytotoxicity. Antineuroblastoma activity will be monitored using standard radiographic & bone marrow studies, as well as RT-PCR for measurement of minimal residual disease in blood & bone marrow. Phase II treatment schema for patients in 1st CR/VGPR or >2nd CR/VGPR will be the same for the vaccine as in phase I except OPT-821 will be given at a fixed dose of 150 mcg/m2.
Biological: oral β-glucan — Phase II Patients will be randomized to starting oral β-glucan (40 mg/kg/day) in week 1 or in week 6.

SUMMARY:
In the first part of this study we found the highest dose of the vaccine that did not have too many side effects. We are now trying to find out what effects the vaccine has when given at the same dose to all patients. The main treatment in this protocol is a vaccine. It is called a " bivalent vaccine" which means it has 2 antigens. An antigen is a specific protein on the surface of a cell. The antigens are called GD2L and GD3L.

We want the vaccine to cause the patient's immune system to make antibodies against the antigens. Antibodies are made by the body to attack cancer (and to fight infections). If the patient can make antibodies against the 2 antigens in the vaccine, those antibodies might also attach to neuroblastoma cells because a lot of each antigen is on neuroblastoma (and very little on other parts of the body). Then, the attached antibodies would attract the patient's white blood cells to kill the neuroblastoma. This protocol also uses β-glucan which is a kind of sugar from yeast. β-glucan is taken by mouth and can help white blood cells kill cancer. The best way to get the body to make antibodies against the 2 antigens is to link each antigen to a protein called KLH (which stands for: keyhole limpet hemocyanin) and to mix them with a substance called QS-21. But it is hard to get enough QS-21 so we are using an identical substance called OPT-821, which we can get easily in large amounts for use in patients.

DETAILED DESCRIPTION:
The phase II treatment schema for patients in 1st CR or ≥ 2nd CR will be the same for the vaccine as in phase I except OPT-821 will be given at a fixed dose of 150 mcg/ m^2 and with no DLT assessment. Patients will be randomized to starting oral β-glucan in week 1 or in week 6.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neuroblastoma (NB) as defined by international criteria,[104] i.e., histopathology (confirmed by the MSKCC Department of Pathology) or bone marrow metastases plus high urine catecholamine levels.
* High-risk NB as defined by risk-related treatment guidelines and the International NB Staging System,[104] i.e., stage 4 with MYCN amplification (any age) stage 4 >18 months old.
* High-risk NB (as defined above) and in 1) first CR at 6 ≥ months from initiation of immunotherapy using anti-GD2 antibody, or 2) second or subsequent remission. Remission is defined as complete (CR) remission, according to the International Neuroblastoma Response Criteria.[104] Urine catecholamine levels are no longer taken into consideration when staging.
* Absolute lymphocyte count ≥ 500/mcl and absolute neutrophil count ≥ 500/mcl.
* Patients with grade 3 toxicities or less using the Common Toxicity Criteria (Version 3.0) developed by the National Cancer Institute of the USA (CTCAE v3.0) related to cardiac, neurological, pulmonary, renal, hepatic or gastrointestinal function as determined by blood tests or physical exam.
* ALT, AST and Alkaline Phosphatase ≤ 2.5 times the upper limit of normal
* Prior treatment with other immunotherapy, including antibodies, is allowed
* ≥ 3 weeks and no more than 6 months (<180 days) between completion of systemic therapy and 1st vaccination.
* Patients previously enrolled on this trial are eligible for repeat enrollment but will be assigned to treatment as per the control arm (Group 1) and will not be included in the biostatistical analyses.
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* History of allergy to KLH, QS-21, OPT-821, or glucan.
* Active life-threatening infection.
* Inability to comply with protocol requirements.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 374 (Actual)
Dates: Start 2009-05-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
To determine the maximally tolerated dose of OPT-821 in a vaccine containing two antigens abundantly expressed on neuroblastoma. (PHASE I) | 2 years
To assess anti-NB activity of the bivalent vaccine plus oral β-glucan in patients who are enrolled with evidence of minimal residual disease (MRD) by molecular biological testing of bone marrow. (PHASE II) | 2 years
To prove the adjuvant effect of oral beta-glucan on anti-GD2 antibody titer among patients who are in first or second (or later) complete | 2 years

SECONDARY OUTCOMES:
To obtain preliminary data on whether subcutaneous administration of the bivalent vaccine produces an immune response directed against the target antigens in patients with high-risk neuroblastoma. (PHASE I) | 2 years
To obtain preliminary data on the anti-neuroblastoma activity of the bivalent vaccine plus oral β-glucan in patients, including measuring the molecular response in blood and bone marrow. (PHASE I) | 2 years
To obtain data on the immune response directed against the target NB-associated antigens in patients as induced by the subcutaneous administration of the bivalent vaccine. (PHASE II) | 2 years
To assess FcRIIa, FcRIIIa, CR3 and CD18 gene polymorphism of leukocytes (effector cells), with a view towards a possible association with outcome. (PHASE II) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Cheung IY, Mauguen A, Modak S, Ragupathi G, Basu EM, Roberts SS, Kushner BH, Cheung NK. Effect of Oral beta-Glucan on Antibody Response to Ganglioside Vaccine in Patients With High-Risk Neuroblastoma: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2023 Feb 1;9(2):242-250. doi: 10.1001/jamaoncol.2022.5999. PMID 36547975
- [Derived] Cheung IY, Cheung NV, Modak S, Mauguen A, Feng Y, Basu E, Roberts SS, Ragupathi G, Kushner BH. Survival Impact of Anti-GD2 Antibody Response in a Phase II Ganglioside Vaccine Trial Among Patients With High-Risk Neuroblastoma With Prior Disease Progression. J Clin Oncol. 2021 Jan 20;39(3):215-226. doi: 10.1200/JCO.20.01892. Epub 2020 Dec 16. PMID 33326254
- [Derived] Kushner BH, Cheung IY, Modak S, Kramer K, Ragupathi G, Cheung NK. Phase I trial of a bivalent gangliosides vaccine in combination with beta-glucan for high-risk neuroblastoma in second or later remission. Clin Cancer Res. 2014 Mar 1;20(5):1375-82. doi: 10.1158/1078-0432.CCR-13-1012. Epub 2014 Feb 11. PMID 24520094
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm